CLINICAL TRIAL: NCT05219058
Title: REMACS - Understanding the Impact of Perineal Reconstruction After Extended MArgin Cancer Surgery on Longer-term Quality of Life, Morbidity and Health Economic Outcomes - a Prospective Longitudinal Cohort Study
Brief Title: Reconstruction in Extended MArgin Cancer Surgery
Acronym: REMACS
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Salisbury NHS Foundation Trust (Other Government); University of Southampton (Other); Dorset County Hospital NHS Foundation Trust (Other Government); The Leeds Teaching Hospitals NHS Trust (Other); Mid Yorkshire Teaching NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospitals Dorset NHS Foundation Trust (Other Government); Somerset NHS Foundation Trust (Other); Swansea Bay University Health Board (Other); Portsmouth Hospitals NHS Trust (Other Government); Hampshire Hospitals NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Sussex Partnership NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); NHS Greater Glasgow and Clyde (Other); The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM OSUR0001
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-07

CONDITIONS: Surgery--Complications; Pelvic Cancer; Abdominal Cancer; Quality of Life
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients undergoing abdominoperineal excision: Abdominoperineal excision alone consists of removing only the rectum and anus
  Interventions: Procedure: Biological mesh reconstruction; Procedure: Myocutaneous flap reconstruction; Procedure: Primary closure reconstruction
- Patient undergoing infralevator pelvic exenteration: Anterior pelvic exenteration includes resection of the structures of the anterior pelvis, namely the bladder, urethra and inner reproductive organs.
  Posterior pelvic exenteration comprises resection of the structures of the posterior pelvic cavity with reproductive organs and rectum, with or without the anal canal.
  Lateral compartment excision describes the resection of pelvic sidewall structures, such as the iliac vessels, piriformis and obturator internus muscles, and ischium, along with sacrotuberous and sacrospinous ligaments.
  Total pelvic exenteration entails removal of the bladder, urethra, inner reproductive organs, rectum, and anus with their muscles and ligaments.
  An infralevator pelvic exenteration includes the removal of the anus with their muscles and ligaments.
  Interventions: Procedure: Biological mesh reconstruction; Procedure: Myocutaneous flap reconstruction; Procedure: Primary closure reconstruction

INTERVENTIONS:
Procedure: Biological mesh reconstruction — Patients receiving biological mesh of any kind or position as part of their reconstruction during surgery.
Procedure: Myocutaneous flap reconstruction — Patients receiving a myocutaneous flap of any kind as part of their reconstruction during surgery.
Procedure: Primary closure reconstruction — Patients receiving primary closure only using any suture material or technique as part of their reconstruction during surgery.

SUMMARY:
Advanced pelvic cancers are uncommon, with treatment being challenging. Around 4000 patients every year need treatment in the UK. Cancers can involve multiple organs and often need radiotherapy and chemotherapy before surgery. Surgery usually requires removal of multiple pelvic organs, including muscles, bone, and skin around the anus (the perineum). This can lead to complications relating to both the empty pelvis syndrome and closure of the perineal defect.

Reconstruction is challenging, with frequently occurring complications, reducing speed of recovery and quality of life. This study investigates complication frequency, quality of life and expenses following different reconstruction techniques. The investigators hope to improve patient and doctor decision-making in this area and find the best methods of reconstruction to improve outcomes.

REMACS has three work packages:

1. Maintenance of a database of patients undergoing colorectal surgery at Southampton and Salisbury Hospitals, including those undergoing extra-levator abdominoperineal excision and pelvic exenteration. This includes all routinely collected clinical data, imaging, health resource use, and patient reported outcome measures.
2. A collaborative national prospective cohort study investigating morbidity, health resource use, longitudinal quality of life outcomes (EORTC QLQ-C30 and disease-specific modules) and quality adjusted life years. The investigators will also assess financial toxicity using the comprehensive score for financial toxicity.
3. A qualitative study using semi-structured interviews to undertake a more complex evaluation of quality of life and patient experiences in patients that have recovered from their surgeries.

The last two work packages have now been funded by an NIHR Research for Patient Benefit Grant

DETAILED DESCRIPTION:
This is an observational multicentre retrospective and prospective cohort study, and a qualitative study. The project will have three working packages:

* Work package 1 - maintenance of a colorectal surgery database
* Work package 2 - prospective collaborative national UK study
* Work package 3 - qualitative analysis with semi-structured interviews

WORK PACKAGE 1 - COLORECTAL SURGERY DATABASE:

Data collected includes:

* Basic demographic information
* Co-morbidities at time of surgery
* Other cancer treatments
* Final cancer staging and diagnosis
* Type of procedure
* Methods of reconstruction
* Use of healthcare resource: (theatre time, surgical teams, use of consumables, index operation intensive care stay, total length of stay, planned or emergency readmissions, use of imaging for complications, re-interventions, and outpatient clinic use).
* Morbidity - empty pelvis syndrome complications with collation of all complications that occurred summarised into: (the highest Clavien-Dindo (CD) score, and the comprehensive complication index by accumulating CD graded complications that a patient has as a result of their surgery.
* Survival: overall and disease-free survival
* Patient reported outcome measures

Any other routinely collected clinical data will be included. Of particular mention we will include and analyse Cardiopulmonary exercise testing data, data derived from the perioperative medicine screening and assessment, data derived from prehabilitation, radiomic data e.g. muscle/fat structure and function derived from CT, MRI or PET-CT.

WORK PACKAGE 2 - PROSPECTIVE COLLABORATIVE STUDY:

Abdominoperineal excision and pelvic exenteration can be used in a wide range of cancer types, and in the case of pelvic exenteration can be used to manage both recurrent and primary cancers. The principal PROM used will be the EORTC QLQ-C30 with its modular questionnaires giving additional insight into disease-specific quality of life.

All amendments have been made in line with NIHR RfPB funding received in November 2024.

Patients will be recruited once a decision to undertake abdominoperineal excision or pelvic exenteration surgery has taken place. Participants will be sent a participant information sheet which will include the dates of when participants can expect follow up telephone calls, with information on how to contact the study team to change these should participants wish to. Once consented participants will undergo the following PROMs as part of their baseline questionnaire:

* EORTC QLQ-C30 with specific cancer-type modules
* EQ-5D-5L
* LRRC QoL
* Decision Regret
* Comprehensive Score for Financial Toxicity (COST), financial status questionnaire (non-validated) and Patient employment status questionnaires.

The investigators anticipate that participants will be able to self-assess the above PROMs on a paper printed form, however a member of the research team will be available to support the participant if required.

Clinical information will also be collected pre-operatively, including: demographic information, co-morbidities, cancer staging, and previous cancer treatments. Patients will be given copies of the follow up questionnaires at this time so participants have them as a reference when completing follow up questionnaires. Patients can opt for either email or telephone follow up for quality of life, if opting for email REDCap study will automatically send out emails based on the date of surgery.

The patient will then undergo their surgery with method of reconstruction at the discretion of the operating surgeon(s).

Following the index admission researchers will enter details on the hospital stay:

* Type of procedure
* Methods of reconstruction
* Theatre time
* Theatre teams
* Use of consumables
* Length of intensive care and hospital stay
* Use of imaging for complications
* Re-interventions for complications
* Discharge destination following index admission
* Final cancer staging and other pathological outcomes.
* Perineal and empty pelvis morbidity, and overall Clavien-Dindo and Comprehensive Complication Index
* NHS healthcare utilisation costs
* If applicable survival and cause of death

At 3 months post-operatively questionnaires will be repeated over the telephone including:

* EORTC QLQ-C30 with cancer-specific module
* EQ-5D-5L
* LRRC QoL
* Decision Regret
* Comprehensive Score for Financial Toxicity (COST), Patient reported heath resource utilisation and NHS healthcare utilisation costs.

At this same time point researchers will review routinely collected clinical data and use of in-hospital health resources to include:

* In-hospital health resource use: planned or emergency re-admissions, use of imaging to investigate complications, re-interventions (surgical and radiological), planned or unplanned outpatient visits.
* Longitudinal CCI scores updated, and if applicable an increase in CD if a more severe complication develops.
* If applicable cancer recurrence, survival and cause of death will be recorded.

Patients will be emailed or telephoned on the date specified on their participant information sheet, however if this time is not convenient then a better time will be arranged with the patient. If participants do not respond to the email or first telephone call then the investigators will make a further three separate attempts to contact the patient. If there is still no response participants will be deemed lost to the study.

This follow up process will be repeated again at 6 months and 12 months. At the 12 month time point the investigators will ask patients additional questions on their use of health care resources and their current financial status, to include:

* Use of community health resource use due to complications including: GP appointments and nursing home care days required for recovery from surgery.
* Use of healthcare resources at hospitals other than the treating hospital - clinic appointments and admissions

At the end of this time the patient will have completed the study.

WORK PACKAGE 3 - QUALITATIVE STUDY:

The qualitative study will recruit patients from work packages 1 and 2. The investigators will invite 30 purposefully sampled patients that are 3 months following their surgery. Suitable patients will be contacted with a posted participant information sheet and a telephone follow up call to allow participants to ask questions about the study. Following informed consent semi-structured interviews will take place with semi-structured open questions to guide the discussions.

Interviews will be recorded on an encrypted audiorecorder and then transcribed. The investigators will initially undertake three pilot interviews to review that the semi-structured interview schedule is adequate to fully explore our objectives and to obtain good quality interview transcripts for analysis. These pilot interviews once completed will be reviewed by the research team. The semi-structured interview schedule questions may be changed if the interviews are of poor quality, pilot interviews demonstrate new insights from participants that suggest fruitful lines of enquiry, or inconsistencies that require further exploration. If subsequent interviews are very different than the pilot interviews following these changes, then these early interviews will not be included in the qualitative analysis and additional patients will be recruited.

Patients recruited at 3-months following surgery will be offered a repeat interview at 12-months following their surgery

DATA ANALYSIS PLAN:

Statistical analysis:

The investigators will be collecting data on the timepoints as described above. Continuous data will be will be summarised using descriptive statistics (mean, median, standard deviation, lower and upper quartiles). Categorical data will be summarised using counts and percentages.

As studies are non-randomised, the investigators will utilise regression models and principal component analysis to adjust for confounding in this observational study.

In order to obtain our outcomes a brief summary of analyses is below.

Work package 1 (Colorectal Database):

Primary analysis:

- Frequency of morbidity relating to the empty pelvis syndrome and perineal wound will be compared for different types of perineal reconstruction will be analysed using multiple linear regression.

Secondary analysis:

* Overall morbidity will be obtained using highest CD scores for different methods of perineal reconstruction analysed using multiple linear regression.
* Disease free and overall survival will be analysed using Kaplan-Meier curves and log rank tests with a multivariate Cox regression hazard model to identify factors independently associated with survival, including method of reconstruction.

Exploratory analysis:

* Other factors including age, gender, BMI, final staging, co-morbidities, type of operation, neoadjuvant chemoradiotherapy and use of intra-operative electron radiotherapy will be included in the analysis
* Other outcomes including primary operation time, lengths of stay, and readmissions will be explored

Work package 2 (prospective study):

Primary and secondary analysis:

* Patient reported outcome measures will be analysed using regression models, including linear mixed-effects models for repeat measures and adjusted analyses.
* The same clinical data fields will be collected as per work package 1, the analysis above repeated with exploratory analysis to find factors that are independently significantly associated with changes in the PROMs.

Health economic analysis:

Work package 1 (retrospective study):

The investigators will collect data on use of hospital healthcare resources in each patient group. The investigators will collect resource use for each parameter required for each patient. The investigators will then undertake costing using a micro-costing approach and health resource group costing for each parameter. Applying costs to each parameter will use a combination of manufacturer prices for consumables, National Cost Collection for the NHS, National Schedule of NHS Costs, NHS National Tariff and the Unit Costs of Health and Social Care from the Personal Social Services Research Unit. The investigators will then report overall costs associated with different methods of perineal reconstruction and the cost of complications that were encountered.

Work package 2 (prospective study):

The investigators will collect hospital healthcare resource use data prospectively and apply micro-costing to these parameters in the same way as per work package 1 for each patient and their method of reconstruction. The investigators will also ask patients to provide us with use of community healthcare resources as a result of their surgery, data for which the investigators will not be able to obtain from their clinical notes. Participants will receive EQ-5D-5L and EORTC QLQ-C30 questionnaires at baseline, 3 months, 6 months and 12 months. From these responses the investigators will map onto EQ-5D-3L in order to reduce the overall number of questionnaires patients are undertaking in our study. This will allow us to plot EQ-5D-3L responses for different methods of reconstruction and plot the area under the curve. Within the trial time a health economic model would be built which would follow the NICE reference case and ISPOR Task Force guidelines on health economic analysis. This will enable us to present Quality Adjusted Life Years and incremental cost-effective ratios for the different methods of perineal reconstruction.

Qualitative analysis:

Audio transcription will be transcribed verbatim, checked against the recording and anonymised. Data will be uploaded to NVivo for data management.

Preliminary summaries will be written after each interview to identify emerging themes to follow-up discussions. The follow-up interview will ask patients to reflect on the content of their previous interview and discuss any changes.

Longitudinal interview analyses will use constant comparative methods from grounded theory and data coded using NVivo's framework matrix facility to examine themes longitudinally, enabling comparisons within each case and across cases, focusing on changes over time. The stages of data analysis, drawing on longitudinal comparisons, will include:

1. Initial reading: Review interview data.
2. Preliminary coding: Two researchers code the data.
3. Team meeting: Discuss and refine codes with wider research/PPI team.
4. Individual Case Coding: Code all interview data for each participant.
5. Categorising Codes: Group codes into categories for each case.
6. Longitudinal comparisons: Within case and category comparisons focussing on changes over time.
7. Focused coding: Examine categories in relation to emerging concepts and phases.
8. Discussion on Themes: PPI co-led focus group discussions of final themes.
9. Development and Dissemination: Report write up are dissemination.

Based on an iterative process, emerging themes will be used to develop explanatory accounts. Analysis will draw on sociological perspectives of illness adaptation, recovery and self-management in addition to psychological theories of individual behaviour change.

All qualitative and quantitative data will inform 3 patient focus groups, where PPI and charity collaborators along with 5 newly trained PPI members will discuss data analyses from a patient perspective, contributing to initial discussions around developing a patient decision aid.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 or older
* Patients that have undergone pelvic exenteration or abdominoperineal excision at participating sites, at any time, that have complete data (work package 1 - Colorectal Surgery Database)
* Patients undergoing pelvic exenteration or abdominoperineal excision at participating sites (work package 2 - prospective study)
* Patients that have already had pelvic exenteration or abdominoperineal resection that can speak English (work package 3 - mixed-methods study)

Exclusion Criteria:

* Patients eligible for, but that are unfit, decline or are not offered abdominoperineal excision or pelvic exenteration surgery
* Patients that undergo surgery by an intersphincteric abdominoperineal resection approach
* Patients that are unable to complete the questionnaire over the telephone or online with a researcher
* Patients unable or unwilling to provide informed consent
* Patients that are prisoners in the custody of HM Prison Service or who are offenders supervised by the probation service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients undergoing abdominoperineal excision or pelvic exenteration for malignancies at thirteen hospitals in England.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Work package 1 | Data collection from prospectively maintained databases over 10 years
  Morbidity for patients undergoing perineal reconstruction following abdominoperineal excision or pelvic exenteration, established by documenting empty pelvis syndrome complications and overall Clavien Dindo scores
Work package 2 | 12 months
  Establishing quality of life in patients undergoing perineal reconstruction with for abdominoperineal excision and pelvic exenteration using The Global European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Scores. Note Global EORTC QLQ-C30 Score ranges from 0 - 100, with a higher score indicating a higher quality of life.
Work package 3 | 3 and 12 months post surgery
  Undertake qualitative analysis from patients' accounts of their experiences in semi-structured interview, in order to complete a more complex evaluation of quality of life after pelvic exenteration and abdominoperineal resection.

SECONDARY OUTCOMES:
Work package 1 | Retrospective data collection over 10 years
  Patient overall and disease-free survival relating to perineal reconstruction.
Work package 1 | Retrospective data collection over 10 years
  Overall costs of perineal reconstructions and the complications that occurred as a result.
Work package 2 | 12 months
  Longitudinal quality of life data (via The Global European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)) in patients undergoing abdominoperineal excision or pelvic exenteration, including disease specific quality of life modules, at 3-months, 6-months and 12-months post-surgery.
  Note that EORTC QLQ-C30 includes scores across functional scales and symptom scales / items, all scores are from 0 to 100, a higher score indicating a higher response level.
Work package 2 | 12 months
  EQ-5D-5L(https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-5l/) will be measured before surgery and at 3,6,12-months after surgery. This is a validated, NICE recommended measure of QoL encompassing 5 domains: mobility, self-care, usual activity, pain/discomfort and anxiety/depression
Work package 2 | 12 months
  Decision-Regret questionnaire(66) is a validated 5-item scale measuring patient treatment-related decisions before surgery and at 3,6,12-months after surgery.
Work package 2 | 12 months
  Incidence of developing complications relating to perineal reconstruction as measured by Clavien Dindo (CD) and Comprehensive Complication Index (CCI) scores at 3-months, 6-months and 12-months post-surgery.
  The EPS dataset is an international Delphi-derived, core outcome dataset specifically assessing morbidity after extended margin cancer surgery and perineal reconstruction.
  Note CD is scored from 0 - 5, with worsening severity of complications with an increasing score; CCI is scored from 0 - 100 with worsening morbidity with a higher score.
Work package 2 | 12 months
  LRRC-QoL will be measured before surgery and at 3,6,12-months after surgery. It is a validated, locally recurrent rectal cancer patient-reported outcome. It consists of 9 multi-item scales(healthcare services, psychological impact, pain, urostomy-related symptoms, lower limb symptoms, stoma, sexual interest and urinary symptoms) and 3 single-item scales tailored for recurrent cancers.
Work Package 2 | 12 months
  A comparison of costs and benefits, with financial toxicity measurements evaluated by the COST questionnaire measured before surgery and at 3,6,12-months.
  Quality-adjusted life years gained assessed using EQ-5D-5L(similar EQ-5D timepoints above)
  Healthcare resource use data will be collected, and unit costs from the National Schedule of NHS Costs will be used to cost resource use over the 12 months after surgery
Work Package 2 | 24 months
  Overall and disease-free survival at 12-months after surgery
Work package 3 | 3 and 12 months after surgery
  Present main themes arising from patients' experiences undergoing different methods of perineal reconstruction to demonstrate where these experiences are similar and where there are disparities.

CONTACTS AND LOCATIONS:
Overall Officials: Kashuf Khan, MBBS MRCS, Principal Investigator — University Hospitals Southampton
Locations (18):
- United Kingdom (18):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Salisbury NHS Foundation Trust, Salisbury, Wiltshire
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Royal Devon University Healthcare NHS Foundation Trust, Cornwell
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - London North West University Healthcare NHS Trust, London
  - Manchester University NHS Foundation Trus, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - University Hospitals Dorset NHS Foundation Trust, Poole
  - Portsmouth Hospitals University NHS Foundation Trust, Portsmouth
  - Swansea Bay University Health Board NHS Wales, Swansea
  - Mid-Yorkshire Hospitals NHS Trust, Wakefield
  - Hampshire Hospitals NHS Foundation Trust, Winchester
  - Somerset NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: Undecided